CLINICAL TRIAL: NCT05315635
Title: Substance Use and Eating Disorders : Food Craving and Addiction Transfer
Acronym: SUED
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-A00126-37
Record Dates: First submitted 2022-03-04; First posted 2022-04-07 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Substance Use Disorders; Eating Disorders
Keywords: Substance Use Disorders; Eating Disorders; Food craving; Addiction transfer; Addiction; Craving
MeSH Terms: conditions — Substance-Related Disorders; Feeding and Eating Disorders; Behavior, Addictive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Epidemiology: Inpatients who initiate treatment for a substance use disorder (SUD) will have to complete self-questionnaires, a clinical psychiatric assessment (MINI) and a cognitive assessment (MoCA).
  These participants will be assessed at admission in addiction unit and at discharge, 3 weeks after withdrawal.
  Outpatients who begin treatment for an eating disorder (ED) will have to complete self-questionnaires and a clinical psychiatric assessment (MINI) at the beginning of the outpatient treatment program
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients treated for substance use disorders and patients treated for eating disorders will have to complete self-questionnaires and a clinical psychiatric (MINI) at the inclusion.
  Patients suffering from substance use disorder will be assessed 3 weeks after inclusion.
  Questionnaires are :
  * Modified Yale Food Addiction (mYFAS 2.0) and Impulsive Behavior Scale (UPPS-P)
  * Trait Meta-Mood Scale (TMMS), Hospital Anxiety and Depression Scale (HADs), Emotional Appetite Questionnaire (EMAQ), Perceived Stress Scale (PSS-10), Multidimensional Assessment of Interoceptive Awareness (MAIA) and Five Facet Mindfulness Questionnaire (FFMQ)
  * Mini International Neuropsychiatric Interview (MINI), Eating Disorder Examination-Questionnaire (EDE-Q), Rosenberg's Self Esteem (RSE) and Ruminative Response Scale for Eating disorders (RRS-ED)
  * Pittsburgh Sleep Quality Index (PSQI) and Montreal Cognitive Assessment (MoCA)

SUMMARY:
Substance Use Disorder (SUD) and Eating Disorders (ED) are severe and persistent disturbances that are associated with significant harm. These two disorders have many clinical similarities, including craving and behavioral loss of control. Recently, craving for food has been described in newly abstinent patients with SUD. the aim of the study is to verify the hypothesis of addiction transfer based on common neurobiological mechanisms between substance craving and food craving, that postulates that food craving would correspond to an attempt to regulate substance craving (or vice versa).

DETAILED DESCRIPTION:
The knowledge of existence of common addictive, neurobiological and clinical processes between substance use disorders and eating disorders has been a promising approach for a better understanding of the factors involved in the emergence and maintenance of these disorders. Several studies have shown that increased palatable food with high sugar or fat content causes brain neurochemistry changes similar to those observed after use of addictive drugs. Clinical and behavioral similarities concerning craving, loss of control and use as a coping strategy have also been highlighted. Craving is considered as a clinical marker of addiction and a potent predictor of relapse vulnerability. In substance addiction, the link between craving, use and relapse has been previously demonstrated in experimental and daily life studies. The main objective of this study is to examine the hypothesis of addiction transfer between Substance Use Disorders and Eating Disorders, according to which food craving for palatable foods would correspond to an attempt to regulate substance craving or vice versa. One assumption is that food intake could be used to alleviate craving for substances in patients hospitalized for substance use disorder. The secondary objective is to explore psychopathological, addictive, and medical similarities between substance use disorder and eating disorder participants. Included patients (group 1: substance use disorder participants and group 2: eating disorder) will be asked to answer different self-questionnaires, as well as a clinical psychiatric (MINI) and cognitive (MoCA) assessment.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnostic criteria for substance use disorder/behavioral addiction (gambling) or an eating disorder (Anorexia nervosa, Bulimia nervosa or Hyperphagia access).
* Begin treatment in addiction complex care unit, located in inter-hospital unit Charles Perrens Hospital and Bordeaux University Hospital
* Non-opposition formulated

Exclusion Criteria:

* Severely impaired physical and/or mental health that, according to the investigator, may affect the participant's compliance with the study and understanding of assessment tools
* Trouble in understanding/writing French
* Hospitalization for less than 3-weeks for patients with substance use disorders or behavioral addiction (gambling)
* Individuals participating in another study that includes an ongoing exclusion period.
* Be under guardianship
* Pregnant and/or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnostic and Statistical Manual (DSM)-5 diagnostic criteria for substance use disorder/behavioral addiction (gambling) or DSM-5 diagnostic criteria for eating disorders (Anorexia nervosa, Bulimia nervosa, Hyperphagia access)
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Craving for substance | At the inclusion
  Measurement of craving for substances by Visual Analogue Scale (VAS) - from 0 (no desire at all) to 10 (very much in demand) / higher scores mean a worse outcome
Craving for substance | At week-3
  Measurement of craving for substances by Visual Analogue Scale (VAS) - from 0 (no desire at all) to 10 (very much in demand) / higher scores mean a worse outcome
Craving for food | At the inclusion
  Measurement of food craving by Food Cravings Questionnaire-Trait-Reduced (FCQ-Tr) - from NEVER to ALLWAYS / higher scores mean a worse or better outcome, depending of the question

SECONDARY OUTCOMES:
Identify common determinants of food craving in patients suffering from ED | At inclusion
  Questionnaires for Addictive characteristics : Modified Yale Food Addiction
Identify common determinants of food craving in patients suffering from ED & SUD - Addictive characteristics : | At inclusion
  Impulsive Behavior Scale 4-point Likert scale: 1 (Agree Strongly), 2 (Agree Some), 3 (Disagree Some), and 4 (Disagree Strongly)
Identify common determinants of food craving in patients suffering from ED & SUD - Emotional characteristics | At inclusion
  Trait Meta-Mood Scale from NOT AT ALL AGREE to TOTALLY AGREE / higher scores mean a worse or better outcome, depending of the question
Identify common determinants of food craving in patients suffering from ED & SUD - Psychopathological and cognitive characteristics | At inclusion
  Eating Disorder Examination-Questionnaire, from NEVER to EVERY DAY / higher scores mean a worse or better outcome, depending of the question
Identify Medical characteristics : of food craving in patients suffering from ED - Medical characteristics : | At inclusion
  BMI in kg/m²
Identify Medical characteristics : of food craving in patients suffering from SUD | At inclusion and at week-3
  BMI in kg/m²
Identify cognitive characteristics of food craving in patients suffering from ED | At inclusion
  Pittsburgh Sleep Quality Index (21 self-rated items are combined to form seven "component scores", each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.) Montreal Cognitive Assessment (30-question test - score of 25 and under is considered at-risk of dementia)
Identify cognitive characteristics of food craving in patients suffering from SUD | At inclusion and at week-3
  Pittsburgh Sleep Quality Index (21 self-rated items are combined to form seven "component scores", each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.) Montreal Cognitive Assessment (30-question test - score of 25 and under is considered at-risk of dementia)
Identify addictive characteristics of substances craving in patients suffering from SUD | At week-3 At inclusion and at week-3
  Impulsive Behavior Scale 4-point Likert scale: 1 (Agree Strongly), 2 (Agree Some), 3 (Disagree Some), and 4 (Disagree Strongly)
Identify emotional characteristics of substances craving in patients suffering from SUD | At week-3
  Trait Meta-Mood Scale, from NOT AT ALL AGREE to TOTALLY AGREE / higher scores mean a worse or better outcome, depending of the question
Identify psychopathological characteristics of substances craving in patients suffering from SUD | At week-3
  Eating Disorder Examination-Questionnaire, from NEVER to EVERY DAY / higher scores mean a worse or better outcome, depending of the question

CONTACTS AND LOCATIONS:
Overall Officials: Mélina FATSEAS, Prof, MD, Study Director — Physician
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Bordeaux, Gironde, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Atkinson TJ. Central and peripheral neuroendocrine peptides and signalling in appetite regulation: considerations for obesity pharmacotherapy. Obes Rev. 2008 Mar;9(2):108-20. doi: 10.1111/j.1467-789X.2007.00412.x. PMID 18257752
- [Result] Avena NM, Murray S, Gold MS. Comparing the effects of food restriction and overeating on brain reward systems. Exp Gerontol. 2013 Oct;48(10):1062-7. doi: 10.1016/j.exger.2013.03.006. Epub 2013 Mar 25. PMID 23535488
- [Result] Bydlowski S, Corcos M, Jeammet P, Paterniti S, Berthoz S, Laurier C, Chambry J, Consoli SM. Emotion-processing deficits in eating disorders. Int J Eat Disord. 2005 May;37(4):321-9. doi: 10.1002/eat.20132. PMID 15856501
- [Result] Calero-Elvira A, Krug I, Davis K, Lopez C, Fernandez-Aranda F, Treasure J. Meta-analysis on drugs in people with eating disorders. Eur Eat Disord Rev. 2009 Jul;17(4):243-59. doi: 10.1002/erv.936. PMID 19475697
- [Result] Canan F, Karaca S, Sogucak S, Gecici O, Kuloglu M. Eating disorders and food addiction in men with heroin use disorder: a controlled study. Eat Weight Disord. 2017 Jun;22(2):249-257. doi: 10.1007/s40519-017-0378-9. Epub 2017 Apr 22. PMID 28434177